CLINICAL TRIAL: NCT01777217
Title: A Pilot Study to Assess the Safety and Efficacy of Solifenacin (VESIcare) for Improving Urinary and Bladder Functions in Patients Undergoing Radiation Therapy of the Prostate
Brief Title: VESIcare For Improving OAB Symptoms in Patients Undergoing IGRT of the Prostate
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated
Sponsor: Advanced Research Network (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VESI-12J03
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2014-12

CONDITIONS: Over-Active Bladder
Keywords: Urination Disorder; Overactive Bladder; Prostate Cancer Radiation; Vesicare
MeSH Terms: conditions — Urination Disorders; Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- solifenacin succinate (Active Comparator): Solifenacin succinate, 5mg or 10 mg once daily
  Interventions: Drug: Solifenacin succinate
- Placebo (Placebo Comparator): Drug: Placebo oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solifenacin succinate — IGRT with VESIcare
  Other Names: VESIcare
  Arms: solifenacin succinate
Drug: Placebo — IGRT with placebo
  Other Names: Control
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if Vesicare (Solifenacin succinate) is effective in treating over-active bladder symptoms during radiation therapy of the prostate.

DETAILED DESCRIPTION:
This is a randomized double blind placebo controlled flexible dose 12 week study. Following screening, subjects will receive their first dose of study medication following completion of AUASS questionnaire on the first day of radiation treatment (baseline) and will continue for twelve weeks. Subjects will be started on 5 mg of study medication. The AUASS will be completed at baseline, weeks 4, 8 and 12. A 16 week visit conducted over a phone interview.

ELIGIBILITY:
Inclusion Criteria:

1. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent and privacy language as per HIPAA Authorization for the USA test sites is obtained from subject or legally authorized representative prior to the initiation of this study (including withdrawal of prohibited medication, if applicable)
2. Subject must be an ambulatory male at least 18 years of age.
3. Subject has been diagnosed with prostate carcinoma and has elected to undergo external beam radiation therapy.
4. Subject is willing to complete the American Urology Association Symptom Score (AUASS) Questionnaire.

Exclusion Criteria:

1. Subject has undergone a prostatectomy
2. Subject exhibits symptoms of urinary tract infection.
3. Subject exhibits severe neurologic damage or has undergone prostatectomy.
4. Subject diagnosed with OAB and is being treated with medication for alleviation of OAB symptoms within 12 months prior to the Screening Visit.
5. Subject has evidence of uncontrolled narrow angle glaucoma, urinary or gastric retention, neurogenic bladder; prostatitis, or persistent UTI.
6. Subject exhibits hypersensitivity to Solifenacin succinate, any ingredients, or other anticholinergic agents.
7. Subject has undergone treatment with any investigational drug within 30 days prior to screening procedure.
8. Subject has exhibited history of diagnosed gastrointestinal obstructive disease.
9. Subjects with co-morbid lower urinary tract symptoms (LUTS).
10. Subjects exhibiting clinically significant bladder outflow obstruction (BOO).
11. In the opinion of the Study Investigator, the patient has exhibited prior to the screening or Baseline visit, a clinically significant disease or medical condition that would exclude the subject from participating in the study.
12. Subjects who have received prior pelvic radiation.
13. Subjects with history of severe hepatic impairment.
14. Subjects with history of Congenital or Acquired QT prolongation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Mehta, M.D., Principal Investigator — Century Cancer Centers
Locations (1):
- Century Cancer Center, Houston, Texas, United States

REFERENCES:
- [Background] Kuban DA, Tucker SL, Dong L, Starkschall G, Huang EH, Cheung MR, Lee AK, Pollack A. Long-term results of the M. D. Anderson randomized dose-escalation trial for prostate cancer. Int J Radiat Oncol Biol Phys. 2008 Jan 1;70(1):67-74. doi: 10.1016/j.ijrobp.2007.06.054. Epub 2007 Aug 31. PMID 17765406
- [Background] Ikeda K, Kobayashi S, Suzuki M, Miyata K, Takeuchi M, Yamada T, Honda K. M(3) receptor antagonism by the novel antimuscarinic agent solifenacin in the urinary bladder and salivary gland. Naunyn Schmiedebergs Arch Pharmacol. 2002 Aug;366(2):97-103. doi: 10.1007/s00210-002-0554-x. Epub 2002 Jun 14. PMID 12122494
- [Background] Michalski JM, Purdy JA, Winter K, Roach M 3rd, Vijayakumar S, Sandler HM, Markoe AM, Ritter MA, Russell KJ, Sailer S, Harms WB, Perez CA, Wilder RB, Hanks GE, Cox JD. Preliminary report of toxicity following 3D radiation therapy for prostate cancer on 3DOG/RTOG 9406. Int J Radiat Oncol Biol Phys. 2000 Jan 15;46(2):391-402. doi: 10.1016/s0360-3016(99)00443-5. PMID 10661346
- [Background] Peeters ST, Heemsbergen WD, Koper PC, van Putten WL, Slot A, Dielwart MF, Bonfrer JM, Incrocci L, Lebesque JV. Dose-response in radiotherapy for localized prostate cancer: results of the Dutch multicenter randomized phase III trial comparing 68 Gy of radiotherapy with 78 Gy. J Clin Oncol. 2006 May 1;24(13):1990-6. doi: 10.1200/JCO.2005.05.2530. PMID 16648499
- [Background] Zelefsky MJ, Yamada Y, Fuks Z, Zhang Z, Hunt M, Cahlon O, Park J, Shippy A. Long-term results of conformal radiotherapy for prostate cancer: impact of dose escalation on biochemical tumor control and distant metastases-free survival outcomes. Int J Radiat Oncol Biol Phys. 2008 Jul 15;71(4):1028-33. doi: 10.1016/j.ijrobp.2007.11.066. Epub 2008 Feb 14. PMID 18280056
- [Background] Zietman AL, DeSilvio ML, Slater JD, Rossi CJ Jr, Miller DW, Adams JA, Shipley WU. Comparison of conventional-dose vs high-dose conformal radiation therapy in clinically localized adenocarcinoma of the prostate: a randomized controlled trial. JAMA. 2005 Sep 14;294(10):1233-9. doi: 10.1001/jama.294.10.1233. PMID 16160131
- [Background] Bostwick DG, Burke HB, Djakiew D, Euling S, Ho SM, Landolph J, Morrison H, Sonawane B, Shifflett T, Waters DJ, Timms B. Human prostate cancer risk factors. Cancer. 2004 Nov 15;101(10 Suppl):2371-490. doi: 10.1002/cncr.20408. PMID 15495199

RESULTS

PARTICIPANT FLOW:
Groups:
- Solifenacin Succinate: Solifenacin succinate, 5mg or 10 mg once daily
  Solifenacin succinate
- Placebo: Drug: Placebo oral
  Placebo
Period: Overall Study
Arm/Group | Solifenacin Succinate | Placebo
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Solifenacin Succinate | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (8.74) | 66 (7.57) | 65.25 (7.61)
Age, Categorical [Count of Participants; unit: Participants] — Participant population is >=50
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 2 | 1 | 3
    >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants] — The participant population are all males
  Participants
    Female | 0 | 0 | 0
    Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Study Measured by the American Urology Association Symptom Score Questionnaire (AUASS).
Description: The AUASS score range is 1-7 (mild), 8-19 (moderate) and 20-35 (severe). The AUASS asks 7 questions scored 0-5, the scores are summed for the total score.
Time Frame: baseline and 16 weeks
Measure: Median (Standard Deviation); unit: Scores on a scale
Arm/Group | Solifenacin Succinate | Placebo
Number analyzed (Participants) | 4 | 4
Scores on a scale | 9.4 (4.24) | 6.7 (4.52)

ADVERSE EVENTS:
Arm/Group | Solifenacin Succinate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No